CLINICAL TRIAL: NCT06708156
Title: The Effectiveness and Safety of Two Low-concentration Atropine Sulfate Eye Drops (0.01%/0.02%) for Delaying the Progression of Myopia in Children and Adolescents in a Randomized, Double-blind, Placebo Parallel-controlled, Multicenter, Phase III Clinical Trial
Brief Title: The Effectiveness and Safety of Two Low-concentration Atropine Sulfate Eye Drops (0.01%/0.02%) for Delaying the Pediatric Myopia Progression
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oupushifang Pharmaceutical Technology Co., Ltd. (Other)
Collaborators: Seefunge Pharmaceutical Technology Co., Ltd. (Industry); AUTEK China Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTR20240786; CTR20240786 (Registry Identifier: National Medical Products Administration, NMPA)
Record Dates: First submitted 2024-11-20; First posted 2024-11-27 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Myopia Progression
Keywords: Myopia; Atropine
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking aims to achieve the unpredictability of randomized treatment groups by all parties involved in a clinical trial. To reduce the influence of evaluation bias or other factors, a double-blind experimental design was adopted in this study. Placebo is the auxiliary ingredient of atropine sulfate eye drops, and its specification, color, smell, etc. are consistent with the test drug and do not contain the active ingredient of the test drug. The drug in the experimental group was packaged in the same packaging as the placebo, and blinded according to random numbers to ensure that both the investigator and the subject were masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (0.01% atropine sulfate eye drops) (Active Comparator): 1 drop in each eye, once a day, every night before sleep, gently press the dacryocyst on both sides for about 1 minute.
  Interventions: Drug: Atropine sulfate eye drops 0.01%
- Experimental group (0.02% atropine sulfate eye drops) (Active Comparator): 1 drop in each eye, once a day, every night before sleep, gently press the dacryocyst on both sides for about 1 minute.
  Interventions: Drug: Atropine sulfate eye drops 0.02%
- Control group (placebo eye drops) (Placebo Comparator): 1 drop in each eye, once a day, every night before sleep, gently press the dacryocyst on both sides for about 1 minute.
  Interventions: Drug: Placebo eye drops

INTERVENTIONS:
Drug: Atropine sulfate eye drops 0.01% — Drug: 0.01% atropine sulfate eye drops Dosage form and strength: 0.01% (0.4 mL: 0.04 mg) eye drops Usage: both eyes, 1 drop in each eye, once a day, every night before sleep, gently press the dacryocyst on both sides for about 1 minute.
  Arms: Experimental group (0.01% atropine sulfate eye drops)
Drug: Atropine sulfate eye drops 0.02% — Drug: 0.02% atropine sulfate eye drops Dosage form and strength: 0.02% (0.4 mL: 0.08 mg) eye drops Usage: both eyes, 1 drop in each eye, once a day, every night before sleep, gently press the dacryocyst on both sides for about 1 minute.
  Arms: Experimental group (0.02% atropine sulfate eye drops)
Drug: Placebo eye drops — Drug: placebo eye drops Dosage form and strength: 0.4 mL eye drops Usage: both eyes, 1 drop in each eye, once a day, every night before sleep, gently press the dacryocyst on both sides for about 1 minute.
  Arms: Control group (placebo eye drops)

SUMMARY:
The clinical trial aims to test the effectiveness and safety of two low-dose atropine sulfate eye drops for delaying myopia progression in children and adolescents.

Primary Objective: evaluate the effectiveness of 0.01% and 0.02% atropine sulfate eye drops for 96 weeks compared to placebo in delaying myopia progression in children and adolescents. Secondary Objective: evaluate the safety of two low-concentration atropine sulfate eye drops (0.01%/0.02%) in delaying myopia progression in children and adolescents.

Exploratory Objective:

1. the efficacy and safety of two low-concentration atropine sulfate eye drops (0.01%/0.02%) for 144 weeks.
2. evaluate the rebound effect of two low-concentration atropine sulfate eye drops (0.01%/0.02%) after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. The legal guardian of the subject voluntarily signed the written informed consent, and the subject over 8 years is required to sign the written informed consent voluntarily.
2. Patients with myopia aged 6 to 12 years, including cut-offs.
3. The equivalent spherical refraction ranges from -1.00 D to -4.00 D (automatic optometry under a cycloplegia condition) in both myopia eyes at inclusion screening.
4. The astigmatism of both eyes was ≤ 1.50 D under a cycloplegia condition at inclusion screening.
5. The antimetropia (measured by equivalent spherical refraction) is < 2.00 D at inclusion screening.
6. Able to comply with study requirements, attend all study visits (including telephone visits), and be willing to receive random grouping of atropine treatment or placebo.

Exclusion Criteria:

1. Allergic to this product or its excipients.
2. Suffering from eye diseases that may affect vision (e.g. lens diseases such as cataracts, glaucoma, fundus macular disease, keratopathy, uveitis, retinal detachment, severe vitreous opacity, etc., manifest strabismus, nystagmus, ocular acute inflammatory disease), history of recurrent chronic ocular inflammation, or any other ocular pathology (e.g., angular stenosis, shallow anterior chamber).
3. Intraocular pressure of either eye is > 21 mmHg or <10 mmHg at screening.
4. Use of low-concentration (0.05% and below) atropine sulfate eye drops (including various in-hospital preparations, except for test drugs) and orthokeratology lenses (OK lenses) within 6 months before the screening.
5. Use of other myopia control methods such as instruments (multifocal glasses, progressive multifocal glasses, etc.), medications (the use of cycloplegic agents for examinations such as optometry is allowed), and others (including traditional Chinese medicine, auricular acupuncture, massage, accommodative flippers, red light therapy instrument, etc.) within 3 months before screening.
6. Those who have participated in other clinical trials and received drug or medical device interventions within 3 months before screening.
7. Systemic or topical use of drugs that affect the efficacy evaluation, such as anticholinergics: atropine, pirenzepine, etc., and cholinomimetics: pilocarpine, etc. within 1 week before screening.
8. Combined with severe immune system disease, central nervous system disease, Down syndrome, asthma, cardiopulmonary insufficiency, liver and kidney dysfunction, etc.
9. Surgical intervention (ocular or systemic) within 6 months before screening, or planned surgery during the study.
10. Heart rate sustained (more than 10 minutes) greater than 120 beats/min at screening (after 10 minutes of rest if the ECG shows a heart rate greater than 120 beats per minute, the ECG should be retested 10 minutes later. If the retest result below 120 beats/min, the screening is successful; If the retest result is still >120 beats/min, screening failed).
11. Need for ocular use or systemic oral corticosteroids during the study. Intranasal, inhaled, topical cutaneous, intra-articular, perianal steroids, and short-term oral steroids (i.e., continuous use for < 2 weeks).
12. Other conditions that are considered unsuitable by the investigator.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 606 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effective change from baseline in equivalent spherical refraction at Week 96 visit | At the Week 96 visit
  The inter-group difference in the value of change from baseline in equivalent spherical refraction after 0.01% or 0.02% atropine sulfate eye drops versus placebo under a cycloplegia condition at the Week 96 visit

SECONDARY OUTCOMES:
Effective change from baseline in eye axis length at 24 months | At the Week 96 visit
  Value of change from baseline in eye axis length at 24 months of dosing (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)
Effective change from baseline in refraction at 12 months | At the Week 48 visit
  Change from baseline in refraction (automatic optometric equivalent spherical refraction under a cycloplegia condition) at 12 months (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)
Effective change from baseline in ocular axis length at 12 months | At the Week 48 visit
  Change from baseline in ocular axis length at 12 months of dosing (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)
Progression of refraction ≤0.50 D at 12 months and 24 months and percentage | At the Week 48 and Week 96 visits
  Progression of refraction (automatic optometric equivalent spherical refraction under a cycloplegia condition) ≤0.50 D at 12 months and 24 months (0.02% atropine vs. placebo; 0.01% atropine vs. placebo) and percentage (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)
Progression of refraction ≤0.75D at 12 months and 24 months and percentage | At the Week 48 and Week 96 visits
  Progression of refraction (automatic optometric equivalent spherical refraction under a cycloplegia condition) ≤0.75D at 12 months and 24 months and percentage (0.02% atropine vs placebo; 0.01% atropine vs placebo)
Progression of refraction ≤1.00D at 12 months and 24 months and percentage | At the Week 48 and Week 96 visits
  Progression of refraction (automatic optometric equivalent spherical refraction under a cycloplegia condition) ≤1.00D at 12 months and 24 months (0.02% atropine vs. placebo; 0.01% atropine vs. placebo) and percentage (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)
Progression of refraction >1.00D at 12 months and 24 months and percentage | At the Week 48 and Week 96 visits
  Progression of refraction (automatic optometric equivalent spherical refraction under a cycloplegia condition) >1.00D at 12 months and 24 months of dosing and percentage (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)
Percentage of patients with 30% and 50% reduction in myopia progression at 12 and 24 months | At the Week 48 and Week 96 visits
  Percentage of patients with 30% and 50% reduction in myopia progression at 12 and 24 months of medication compared to control (0.02% atropine versus placebo; 0.01% atropine versus placebo)
Change from baseline in other ocular morphologic measures at 12 months and 24 months | At the Week 48 and Week 96 visits
  Change from baseline in other ocular morphologic measures (e.g., corneal curvature, vitreous chamber depth, choroidal thickness) at 12 months and 24 months of dosing (0.02% atropine vs. placebo; 0.01% atropine vs. placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, Postdoctoral, Principal Investigator — Beijing Tongren Hospital Affiliated to Capital Medical University
Locations (25):
- China (25):
  - Hefei Maternal and Child Health Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First People's Hospital of Zunyi, Zunyi, Guizhou
  - Daqingshi People's Hospital, Daqing, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Weifang Eye Hospital, Weifang, Shandong
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chongqing Aier Eye Hospital, Chongqing
  - Shanghai Eye Disease Prevention and Treatment Center (Shanghai Eye Hospital), Shanghai
  - Tianjin Medical University Eye Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No